CLINICAL TRIAL: NCT01368887
Title: Phase II Study of a Non-Steroidal Novel Treatment for Scalp Psoriasis
Brief Title: Study to Test the Effectiveness of a New Treatment for Scalp Psoriasis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor seeking additional financial support before starting the study
Sponsor: DermiPsor, Ltd. (Industry)
Responsible Party: Shay Marcus, VP Business Development & Marketing, DermiPsor Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DermiPsor 2008-103
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Psoriasis
Keywords: psoriasis; scalp psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): DPS-102
  Interventions: Drug: DPS-102
- 2 (Placebo Comparator): Vehicle
  Interventions: Other: Vehicle / Placebo
- 3 (Active Comparator): Calcipotriol Monotherapy
  Interventions: Drug: Calcipotriol Monotherapy
- 4 (Active Comparator): Nicotinamide Monotherapy
  Interventions: Drug: Nicotinamide Monotherapy

INTERVENTIONS:
Drug: DPS-102 — The patient will apply the treatment twice daily in the morning and at bedtime on the involved area only. The scheduled treatment duration is 12 weeks. Patient to begin treatment on the night of Visit 1.
  Arms: 1
Other: Vehicle / Placebo — The patient will apply the vehicle twice daily in the morning and at bedtime on the involved area only. The scheduled treatment duration is 12 weeks. Patient to begin treatment on the night of Visit 1.
  Arms: 2
Drug: Calcipotriol Monotherapy — The patient will apply the treatment twice daily in the morning and at bedtime on the involved area only. The scheduled treatment duration is 12 weeks. Patient to begin treatment on the night of Visit 1.
  Arms: 3
Drug: Nicotinamide Monotherapy — The patient will apply the treatment twice daily in the morning and at bedtime on the involved area only. The scheduled treatment duration is 12 weeks. Patient to begin treatment on the night of Visit 1.
  Arms: 4

SUMMARY:
The purpose of this study is to test the effectiveness of DermiPsor's DPS-102 (test product) in patients with scalp Psoroasis. The study is also intended to assess the safety of the product.

DETAILED DESCRIPTION:
Psoriasis is a non-contagious skin disorder affecting up to 2% of the world population. It is estimated that 26 million people in the U.S. and Europe suffer from psoriasis. Forty percent (40%) of these suffer from psoriasis of the scalp. Currently, there are three primary modalities for the treatment of psoriasis: topical, phototherapy and systemic treatments. While existing treatments provide varying degrees of relief for this illness, they do not provide a long-term cure. Additionally, there is evidence that some of these existing treatments may cause significant side effect. The purpose of this study is to demonstrate that DermiPsor's DPS-102 (test product) is statistically more effective for the treatment of psoriasis current topical treatment options. It is also intended to assess the safety of DPS-102.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age 18 or older
* Patient with a personal history of scalp psoriasis
* Patient with treatable lesions
* Patient with a TSS score equal or lower than 9.
* Patient with a PGA score equal or lower than 5.
* Patient with a negative urine pregnancy test at inclusion for women of childbearing potential and using an efficient contraceptive (oral contraceptives, IUD, or tubal ligation)
* Patient agreeing to participate to the study and to sign a written informed consent and comply with study requirements.

Exclusion Criteria:

* Patient treated with topical scalp treatment for scalp psoriasis within two weeks prior to the inclusion in the study (corticoids, retinoids, vitamin D derivatives),
* Patient treated with systemic treatment for psoriasis (biologics, methotrexate, cyclosporine, retinoids) within one month prior to the inclusion in the study
* Patient taking systemic niacin or multivitamins within past two weeks
* Patient who start or modify a treatment with beta-blockers within one month prior to the inclusion in the study
* Patient with PEG (Poly Ethylene Glycol) allergy
* Pregnant or breast feeding female or female who do not use contraception,
* Patient with an history of hypersensitivity to Dovonex/Daivonex
* Patient who has participated in a clinical trial within three month prior inclusion,
* Patients on Carbamazepine and Primidione (the clearance of Primidione and Carbamazepine may be reduced with the concomitant use of Nicotinamide)
* Patient who is under guardianship, or unable to understand the information (for linguistic or mental reason), or unwilling to give her/his informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-11 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The Physician's Global Assessment ("PGA") criteria. The PGA involves a 7 point scale (clear, minimal, mild, moderate, severe and very severe) and grading conducted at 0, 2, 4, 8 and 12 weeks. | 12 weeks
  The number of participants at each PGA scale level assessed at 0,2,4,8,and 12 weeks and a comparison of each individual's scale assessments over the 12 week period to assess any changes.

SECONDARY OUTCOMES:
Review of haematology and blood chemistry test results, and any adverse event reports received. | 12 weeks
  Number of participants who experience adverse events and type of adverse event in each case.

CONTACTS AND LOCATIONS:
Overall Officials: Shay Marcus, Study Director — Sponsor / DermiPsor Ltd.; Nelli Konnikov, M.D., Principal Investigator — Veterans Administration (VA) Hospital - Brockton, MA; Nancy Naguib, M.D., Principal Investigator — Brockton VA Hospital; Carolyn Stanger, Principal Investigator — Boston VA Hospital
Locations (2):
- United States (2):
  - Boston VA Hospital, Boston, Massachusetts
  - Brockton VA Hospital, Brockton, Massachusetts